CLINICAL TRIAL: NCT06218186
Title: A Single Arm Quantitative Study Assessing Performance of Wesper Lab as a Tool to Aid in Sleep Apnea Diagnosis in Pediatric Populations
Brief Title: Assessing the Performance of Wesper Lab for Sleep Apnea Diagnosis in Pediatric Populations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wesper Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: WSP-111
Record Dates: First submitted 2024-01-11; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Sleep Apnea; Sleep Apnea Syndromes in Children; Sleep Apnea Syndromes
Keywords: Sleep Apnea; Pediatric Sleep Apnea; Home Sleep Test; Sleep Disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Medical device, single arm. All subjects will be provided with the same medical device (Wesper Lab), a home sleep test.
Masking Description: All studies will be presented on the same viewing and scoring platform. The sleep study readers will be blinded to patient identification and the data collection device for each study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Medical Device: Wesper Lab (Single Arm) (Experimental): Participants already undergoing a prescribed polysomnography (PSG) sleep study for the diagnosis of sleep apnea will be asked to simultaneously wear Wesper Lab, a home sleep test device.
  Interventions: Device: Medical Device: Wesper Lab Home Sleep Test

INTERVENTIONS:
Device: Medical Device: Wesper Lab Home Sleep Test — Wesper Lab is a medical device that is used for the diagnosis of sleep apnea. Wesper lab is composed of two flexible biosensors that adhere to the abdomen and thorax with medical grade adhesive. A FDA approved pulse oximeter is worn on a finger.

SUMMARY:
The goal of this single arm study is to evaluate the effectiveness of Wesper Lab, previously known as TatchSleep Pro, a wireless home sleep test, as a tool to aid in sleep apnea diagnosis as compared to an overnight polysomnography (PSG) evaluation in a pediatric population (subjects 2 to 21 years of age).

The main question[s] it aims to answer are:

* Does Wesper Lab demonstrate agreement with PSG for the calculation of the apnea/hypopnea index (AHI)?
* Does Wesper Lab demonstrate agreement with PFG for the calculation of sleep apnea severity.

Participants that are already undergoing a prescribed PSG for the detection of sleep apnea will be asked to simultaneously wear the Wesper Lab sensors and an FDA approved pulse oximeter.

Researchers will compare the AHI of Wesper Lab to the AHI of the PSG to determine the accuracy of the Wesper Lab device.

This is a single center, single-arm, quantitative study

DETAILED DESCRIPTION:
This is a single center, single-arm, quantitative study evaluating the effectiveness of the Wesper Lab, previously known as TatchSleep Pro, wireless sensors as a tool to aid in sleep apnea diagnosis as compared to an overnight polysomnography (PSG) evaluation in a pediatric population.

Investigators will identify approximately 150 eligible pediatric patients, 50 subjects per subgroup, who have been recommended to receive an overnight PSG for the detection/evaluation of sleep apnea. Subgroups include pediatric patients in the following age ranges: subgroup 1: 2-5 years old, subgroup 2: 6-11 years old, subgroup 3: 12-21 years old.

After informed consent is obtained, a brief sleep-related medical history will be collected including relevant demographics. Females of childbearing potential (12 years or older) will be asked to undergo a urine dipstick pregnancy test to determine their eligibility for inclusion in the study.

Patients will undergo their PSG test while simultaneously wearing 2 Wesper Lab patches and an FDA-cleared pulse oximeter compatible with and connected to the Wesper Lab system for a single night at the clinic. The same make and model of pulse oximeter will be used for all subjects. Patients will be observed overnight by trained sleep technicians who will setup the Wesper Lab device and collect the sleep data via the companion smartphone application.

A follow-up communication will be made with patients within 5 days after the sleep study to assess any adverse events.

Following the data collection, sleep data from PSG and Wesper Lab will be scored by an independent qualified sleep technologist (the primary reader) to yield an analysis of the accuracy of Wesper Lab compared with the PSG signals. At least one and up to two additional readers (secondary readers) will score only the Wesper Lab data to obtain an estimate of inter-rater reliability.

Accuracy of the Wesper Lab device will be demonstrated by comparing the Pearson correlation of Wesper Lab and PSG AHI to a performance goal. The performance goal is based on a meta-analysis of FDA-cleared similar devices. Fisher's transformation and one-sided Z-test will be used to test the hypotheses with a significance level of 0.025. The upper and lower 95% Bland-Altman limits of agreement will be calculated and statistically compared using a Wald test to performance goals based on a meta-analysis of FDA-cleared similar devices. Deming regression will also be presented. The inter-rater reliability of Wesper Lab AHIs will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Be 2 to 21 years of age.
* Have a referral to the study site from a physician to complete an overnight polysomnogram test for sleep apnea detection or follow-up.
* Be willing and able to wear two Wesper Lab patches and an FDA-cleared pulse oximeter in conjunction with a polysomnogram, for a single night.
* If 18 years or older, be able to willingly sign a written informed consent form prior to the initiation of any study procedure. If younger than 18 years of age, have a parent or legal guardian voluntarily willing to sign a written informed consent form prior to the initiation of any study procedures. Adult patients unable to provide written informed consent on their own behalf will not be eligible for the study.

Exclusion Criteria:

* Individuals younger than 2 years of age.
* Individuals older than 21 years of age
* Females 12 years or older who have a positive urine pregnancy test on the day of the study.
* Any known health condition that, in the opinion of the Investigator, would exclude the patient from participating in the study.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Agreement of Wesper Lab with Polysomnography (PSG) for the scoring of the apnea/hypopnea index (AHI). | 8 hours
  The apnea/hypopnea index (AHI) is a measurement of the presence and seventy of sleep apnea. AHI is the average number of apneas and hypopnea per hour of recorded sleep time, as determined by the American Academy of Sleep Medicine.
  The primary outcome measure of this study is to determine there is sufficient agreement between the AHI measured by Wesper Lab with the AHI measured by PSG.

SECONDARY OUTCOMES:
Agreement of Wesper Lab with Polysomnography (PSG) for the calculation of sleep apnea severity. | 8 hours
  The apnea/hypopnea index (AHI) is a measurement of the presence and seventy of sleep apnea. AHI is the average number of apneas and hypopnea per hour of recorded sleep time, as determined by the American Academy of Sleep Medicine.
  Sleep apnea severity is calculated with AHI as determined by the American Academy of Sleep Medicine.
  Normal: AHI = 0 - 4.99 Mild: AHI = 5 - 14.99 Moderate: AHI = 15 - 29.99 Severe: AHI = >30
  The secondary outcome measure is to determine there is sufficient agreement between the sleep apnea severity measured by Wesper Lab with the sleep apnea severity measured by PSG.

CONTACTS AND LOCATIONS:
Overall Officials: German P Digoy, M.D., Principal Investigator — Associate Professor of Otolaryngology, Oklahoma State University Center for Health Sciences
Locations (1):
- Summit Medical Center, Edmond, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Raphelson JR, Ahmed IM, Ancoli-Israel S, Ojile J, Pearson S, Bennett N, Uhles ML, Rohrscheib C, Malhotra A. Evaluation of a novel device to assess obstructive sleep apnea and body position. J Clin Sleep Med. 2023 Sep 1;19(9):1643-1649. doi: 10.5664/jcsm.10644. PMID 37140998
- [Result] Zandieh S, Kirschenbaum MA, Greenberg H, Ancoli-Israel S. Keep it simple: A novel technique for measuring airflow using a wireless patch. Sleep Health. 2023 Feb;9(1):100-107. doi: 10.1016/j.sleh.2022.10.005. Epub 2022 Dec 5. PMID 36473786
- See also: Investigational Device — http://www.wesper.co